CLINICAL TRIAL: NCT01171222
Title: Health Status and Cardiovascular Stress of Veteran Soccer Players
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Prof. Dr. Tim Meyer, Saarland University
Other Study IDs: Saarland University
Record Dates: First submitted 2010-07-22; First posted 2010-07-28 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2010-07

CONDITIONS: Health Status; Stress
Keywords: soccer; prevention; veteran athletes; exercise; Cardiovascular
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- veteran soccer players from Saarland County, Germany

SUMMARY:
This study shall provide missing descriptive data on health status of veteran players and potential preventive effects of soccer at an age of 40 to 60 years. The investigation represents a cross-sectional examination of cardiovascular parameters and metabolic stress induced by training and competition. Additionally, orthopedic and other medical risks are to be revealed, and options should be developed to minimize these risks, e.g. by preventive measures included in training or rule modifications.

DETAILED DESCRIPTION:
Facing the demographic trends in Western societies there is an expected increase in interest in soccer for males between 40 and 60 years. Positive effects of such an activity on health can be suspected based on some studies and analogous conclusions. However, no sufficient database is available yet. Moreover, the range of cardiovascular risk factors or pre-existing diseases for this specific population is not known.

This study shall provide missing descriptive data on health status of veteran players and potential preventive effects of soccer at an age of 40 to 60 years. The investigation represents a cross-sectional examination of cardiovascular parameters and metabolic stress induced by training and competition. Additionally, orthopedic and other medical risks are to be revealed, and options should be developed to minimize these risks, e.g. by preventive measures included in training or rule modifications.

ELIGIBILITY:
Inclusion Criteria:

* Male veteran soccer players aged 40 years and older, who are member of a club veteran team

Exclusion Criteria:

* Diseases or injuries which are contraindications for physical exercise

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: veteran soccer players from Saarland County, Germany
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Descriptive data from medical check up and physiological testing | 6 months
  The investigation represents a cross-sectional examination of cardiovascular parameters and metabolic stress induced by training and competition:
  * resting ECG
  * stress ECG
  * blood sample
  * VO2max
  * visit of training and competition (including the measurement of heart rate and blood lactate)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Meyer, Prof. Dr., Principal Investigator — Universität des Saarlandes
Locations (1):
- Saarland University, Saarbrücken, Saarland, Germany